CLINICAL TRIAL: NCT06050837
Title: Spleen Stiffness as a Measure to Assess the REsponse to β Blocker Therapy (SPARE-B).
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-SPARE-B-01
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: High Risk Esophageal Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
HVPG is the gold standard for measurement of the presence and severity of portal hypertension. Clinically Significant Portal Hypertension (CSPH) is defined as HVPG ≥ 10 mmHg. Reducing the HVPG by use of non-selective beta blockers has been associated with reduced risk of variceal hemorrhage, ascites, SBP and thus has a positive effect on survival. Response to Beta blocker therapy is defined as a reduction of HVPG by 10% or to ≤ 12 mmHg.

HVPG is an invasive method of assessment of portal pressures, with lack of availability at many centres. While non-invasive tests to predict CSPH have been defined, predicting response to beta-blockers non-invasively is an unmet clinical need.

The aim of this study is to use splenic stiffness measurement, a non-invasive test, as a surrogate to assess the response of HVPG to beta blocker therapy.

DETAILED DESCRIPTION:
Aim and Objective: To evaluate change in splenic stiffness measurement as a surrogate for response to non-selective beta blockers in patients with high-risk esophageal varices.

Primary objectives: To evaluate the diagnostic accuracy of change in splenic stiffness to predict HVPG responders to beta-blockers at 4 weeks

- Study population: All patients aged ≥ 18 years and ≤ 70 years presenting to Institute of Liver and Biliary Sciences, New Delhi with high-risk esophageal varices upon presentation and are giving written consent for participation in the study.

* Study design - Single center, Prospective, observational study.
* Study period - 1 year
* Sample size - We are enrolling 130 patients in the study
* Intervention - Carvedilol will be initiated to all patients with high-risk esophageal varices (in the absence of any contraindications) at a dose of 3.125mg BD and titrated to the maximum tolerable dose within 7 days.
* Monitoring and assessment -
* Investigations - performed at Baseline

  1. CBC, RFT, LFT, PT/INR, vWF-Ag, HbA1c
  2. Collagen markers: Procollagen 3 peptide, tissue inhibitor of matrix metalloproteinase 1, Hyaluronic acid
  3. ECG
  4. 2D Echocardiography
  5. CECT Whole Abdomen
  6. Splenic stiffness measurement
  7. Liver stiffness measurement
  8. Upper GI endoscopy
  9. HVPG
* Investigations - performed at 1 month of maximum tolerable dose of Carvedilol

  1. CBC, RFT, LFT, PT/INR, vWF-Ag
  2. Collagen markers: Procollagen 3 peptide, tissue inhibitor of matrix metalloproteinase 1, Hyaluronic acid
  3. ECG
  4. Splenic stiffness measurement
  5. Liver stiffness measurement
  6. HVPG
* Adverse effects (of carvedilol)

  1. Allergy
  2. Light headedness
  3. Exercise intolerance
  4. Fatigue
  5. Chest tightness

Stopping rule - Development of variceal bleed

Expected outcome of the project:

Change in splenic stiffness will correlates with change in HVPG and can reliably predict response to non-selective beta blockers in patient with high-risk esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Cirrhosis of liver of different etiologies, with evidence of high-risk esophageal varices
3. Alcohol abstinence for 3 months
4. Written informed consent

Exclusion Criteria:

1. Age ≥ 70 years
2. Previous or imminent variceal ligation
3. Non Cirrhotic Portal Hypertension
4. Portal vein, splenic vein thrombosis
5. Porto-systemic shunts > 10 mm
6. Patients already on beta blockers
7. Contraindications to beta blocker therapy :

   1. Heart rate < 50 bpm
   2. Systolic BP < 100 mm Hg
   3. Severe COPD
   4. Atrioventricular block
   5. Known PVD
   6. Poor control of T2DM (HbA1c>9)
8. Technical difficulties for splenic stiffness measurement
9. Cardio-pulmonary disorders
10. Budd Chiari Syndrome
11. Grade 3 ascites
12. Acute Kidney Injury or Chronic Kidney Disease
13. Severely Obese patients (BMI > 40)
14. Pregnant women
15. Advanced HCC
16. Psychiatric Illness
17. Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥ 18 years and ≤ 70 years presenting to Institute of Liver and Biliary Sciences, New Delhi with high-risk esophageal varices upon presentation and are giving written consent for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic accuracy of change in splenic stiffness to predict HVPG responders to beta-blockers at 4 weeks | 4 weeks

SECONDARY OUTCOMES:
Change in Liver stiffness measurement | 4 weeks
Change in Fib-4, Fib-5 | 4 weeks
Change in vWF-antigen, VITRO | 4 weeks
Change in collagen markers - Procollagen 3 peptide, tissue inhibitor of matrix metalloproteinase 1, Hyaluronic acid | 4 weeks
To develop an AI based model to predict HVPG responders to beta blockers | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No